CLINICAL TRIAL: NCT02491359
Title: Carfilzomib for Treatment of Chronic Graft vs. Host Disease
Brief Title: Carfilzomib in Treating Patients With Chronic Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9228; NCI-2015-00809 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9228.00; 9228 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-06-10; First posted 2015-07-08 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carfilzomib) (Experimental): Patients receive carfilzomib IV over approximately 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot phase II trial studies how well carfilzomib works in treating patients with chronic graft-versus-host disease. Chronic graft-versus-host disease is a complication of a donor bone marrow or blood cell transplant, usually occurring more than three months after transplant, in which donor cells damage the host tissue. Carfilzomib may be an effective treatment for chronic graft-versus-host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine proportion of subjects with treatment failure by 6 months of carfilzomib therapy for chronic graft-versus-host disease (GVHD).

SECONDARY OBJECTIVES:

I. Determine 3 month overall (complete + partial), and complete response rate.

II. Determine 6 month overall (complete + partial), and complete response rate.

III. Report overall survival, non-relapse mortality, primary malignancy relapse, failure-free survival, treatment success, and discontinuation of immune suppression at 6 months and 1 year.

IV. Examine functional outcome (2-minute walk test) and patient-reported outcomes (Lee Chronic GVHD Symptom Scale, quality of life [Short Form Health Survey (SF)-36, Functional Assessment of Cancer Therapy Bone Marrow Transplant (FACT-BMT) Questionnaire], Human Activity Profile [HAP]) at study enrollment, 6 months, and 1 year.

V. Study biologic effects of proteasome inhibition.

OUTLINE:

Patients receive carfilzomib intravenously (IV) over approximately 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic GVHD according to National Institutes of Health (NIH) Consensus Criteria

  * May have either classic chronic GVHD or overlap subtype of chronic GVHD
* Failure of at least one prior line of systemic immune suppressive therapy for management of chronic GVHD
* Subject underwent transplantation at least 3 months prior to enrollment
* Anticipated life expectancy >= 6 months
* Alanine aminotransferase (ALT) =< 3.5 times the upper limit of normal, unless due to chronic GVHD
* Bilirubin =< 2 mg/dL, unless due to chronic GVHD
* Absolute neutrophil count (ANC) >= 1.0 × 10^9/L
* Hemoglobin >= 8 g/dL
* Platelet count >= 50 × 10^9/L
* Creatinine clearance (CrCl) >= 15 mL/minute, either measured or calculated
* Signed informed consent in accordance with federal, local, and institutional guidelines
* Females of childbearing potential (FCBP) must agree to a pregnancy test at study enrollment and to practice contraception during the study
* Male subjects must agree to practice contraception during the study

Exclusion Criteria:

* Evidence of recurrent or progressive underlying malignant disease
* Pregnant or lactating females
* Surgery within 21 days prior to enrollment

  * Does not include placement of venous access device, bone marrow biopsy, GVHD diagnostic biopsy, or other routine procedures in chronic GVHD or post-transplantation care
* Uncontrolled infection within 14 days prior to enrollment

  * Infection treated with appropriate antimicrobial therapy and without signs of progression/treatment failure does not constitute an exclusion criterion
* Documented human immunodeficiency virus (HIV) infection
* Active hepatitis B or C infection
* Documented unstable angina or myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or grade 3 conduction system abnormalities (unless subject has a pacemaker), left ventricular ejection fraction (LVEF) < 40%, history of torsade de pointe
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment

  * Sustained systolic blood pressure > 160 or diastolic blood pressure > 100 despite medical therapy; sustained blood sugar > 300 despite medical therapy
  * Chronic hypertension or diabetes on appropriate medical therapy does not constitute an exclusion criterion
* Non-hematologic malignancy within the past 3 years with the exception of:

  * Adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer
  * Carcinoma in situ of the cervix or breast
  * Prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen levels
  * Cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study
* Significant neuropathy per Common Terminology Criteria for Adverse Events (CTCAE) version (ver.) 4.03 or current version (grade 3 and above, or grade 2 with pain) within 14 days prior to enrollment
* History of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
* Contraindication to all available herpes simplex virus (HSV)/varicella prophylactic antiviral drugs
* Pleural effusions requiring thoracentesis, or ascites requiring paracentesis, within 14 days prior to enrollment
* Any other clinically significant medical or psychological disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
* New systemic immune suppressive agent added for the treatment of chronic GVHD within 2 weeks prior to enrollment
* Treatment with a non-Food and Drug Administration (FDA) approved drug in the previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Carfilzomib)
Started | 20
Completed | 4
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [46 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Primary Disease [Count of Participants; unit: Participants]
  Acute leukemia (ALL/AML) | 12
  Chronic leukemia (CML/CLL) | 4
  Lymphoma (NHL/HD) | 2
  Myeloma | 1
  Myeloproliferative neoplasm | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: according to National Cancer Institute CTCAE, version 4.03
Time Frame: Up to 30 days following completion of study treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
participants
  Serious Adverse Events | 8
  Non-Serious Adverse Events | 7

2. Primary Outcome: Probability of Treatment Failure at 6mo
Description: Kaplan-Meier estimate assessed at 6 months for treatment failure, defined as requirement of an additional line of systemic immune-suppressive therapy, recurrent malignancy, or death.
Time Frame: 6 months
Measure: Number; unit: probability of treatment failure
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
probability of treatment failure | 0.4

3. Secondary Outcome: Complete Response Rate
Description: Complete response (CR) at 6 months will be determined by both clinician-defined CR, as well as separately calculated according to the proposed response definitions of the NIH Consensus Conference.
Time Frame: Up to 6 months
Population: Participants who could be evaluated for response (not missing data)
Measure: Number; unit: participants
Groups:
- Response Evaluated by MD; Response Evaluated by NIH: Participants who receive carfilzomib
Arm/Group | Response Evaluated by MD | Response Evaluated by NIH
Number analyzed (Participants) | 16 | 16
participants
  partial response | 5 | 4
  mixed response | 0 | 4
  unchanged | 2 | 1
  progressive | 2 | 0
  failed | 7 | 7

4. Secondary Outcome: Cumulative Incidence of Non-relapse Mortality and Primary Malignancy Relapse
Description: The cumulative incidence of non-relapse mortality (defined as death in the absence of primary malignancy relapse after transplant) and relapse (defined as hematologic relapse or any unplanned intervention to prevent progression of disease in patients with evidence (molecular, cytogenetic, flow cytometric, radiographic) of malignant disease after transplantation) will be estimated from time of study therapy initiation. These will be treated as competing-risk events, and estimated at 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
Participants | 7

5. Secondary Outcome: Probability of Failure-free Survival at 1 Year
Description: Kaplain-Meier estimate assessed at 1 year for failure-free survival, defined as absence of death from any cause, relapse, or addition of secondary immune-suppressive agents.
Time Frame: 1 year
Measure: Number; unit: probability of failure-free survival
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
probability of failure-free survival | .32

6. Secondary Outcome: Impact of Proteasome Inhibition
Description: The biologic impact of proteasome inhibition in the treatment of chronic GVHD will be assessed at baseline, 3 and 6 months. The association between biologic outcome measures and clinical parameters (response, treatment failure, mortality) will be studied.
Time Frame: Up to 6 months
Population: Data were not collected because biologic studies were not performed. Response to study drug too minimal to justify time and expense.
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of Discontinuation of All Systemic Immune-suppressive Therapies
Description: The incidence of complete discontinuation of all systemic immune-suppressive therapies will be determined at 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
Participants | 2

8. Secondary Outcome: Overall Response Rate
Description: Overall response rate (ORR) (complete response + partial response) at 6 months will be determined by both clinician-defined categories of complete response and partial response, as well as separately calculated according to the proposed response definitions of the NIH Consensus Conference.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
participants
  Physician impression ORR | 4
  NIH ORR | 3

9. Secondary Outcome: Probability of Overall Survival at 1 Year
Description: Kaplan-Meier estimate assessed at 1 year for overall survival, defined as absence of death from any cause.
Time Frame: 1 year
Measure: Number; unit: probability of overall survival
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
probability of overall survival | .65

10. Secondary Outcome: Treatment Success
Description: Treatment success will be estimated at 1 year with a composite outcome of complete resolution of all reversible chronic GVHD manifestations, discontinuation of all systemic immune suppressive agents, and freedom from death or primary malignancy relapse after transplant.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
participants | 0

11. Secondary Outcome: Use of Additional Systemic Immune-suppressive Therapies
Description: Addition of therapy after carfilzomib constitutes failure, could occur at any time from baseline to 12mo.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
participants | 13

12. Secondary Outcome: Symptoms as Measured by Patient Self-report--Short Form-36 (SF-36)
Description: SF-36 subscales have min=0 and max=100; results given are actual scores at 12mo, with higher scores indicating higher quality of life.
Time Frame: baseline
Population: Only baseline surveys analyzed. Only 7 patients completed surveys at 6mo, not analyzed due to low number.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
units on a scale
  Norm-based physical functioning | 36 [14.9 to 52.8]
  norm-based role-physical score | 33.6 [17.7 to 54.4]
  norm-based bodily pain score | 41.4 [19.9 to 62.1]
  norm-based general health score | 32.9 [23.4 to 48.2]
  norm-based vitality score | 42.7 [30.2 to 64.6]
  norm-based social functioning | 40.5 [13.2 to 56.8]
  norm-based role-emotional score | 40.3 [17 to 55.9]
  norm-based mental health score | 50 [33.1 to 61.3]
  standardized physical component score | 37 [15.9 to 52.2]
  standardized mental component score | 49 [28.6 to 64.1]

13. Secondary Outcome: Symptoms as Measured by Patient Self-report--Functional Assessment of Chronic Illness Therapy (FACT)
Description: FACT-BMT subscales have various min/max, see below; results given are actual 12mo scores, with higher scores indicating better functioning.
  FACT physical well-being (0-28) FACT social/family well-being (0-28) FACT emotional well-being (0-24) FACT functional well-being (0-28) FACT Bone Marrow Transplant (BMT) subscale (0-40) FACT trial outcome index (0-96) FACT-General (G) (0-108) FACT-BMT total (0-148)
Time Frame: baseline
Population: Only baseline surveys analyzed. Only 7 patients completed surveys at 6mo, not analyzed due to low number.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
units on a scale
  physical well-being | 21.5 [7 to 26]
  social/family well-being | 21.5 [15 to 28]
  emotional well-being | 18.5 [8 to 24]
  functional well-being | 16.5 [5 to 23]
  BMT subscale | 28 [21 to 33.3]
  FACT-G | 72.8 [53 to 98]
  trial outcome index | 65 [39 to 81]
  FACT-BMT total | 101.3 [75 to 131.3]

14. Secondary Outcome: Symptoms as Measured by Patient Self-report--Human Activities Profile (HAP)
Description: HAP subscales have min=0 and max=94; results given are actual 12mo scores, with higher scores indicating better functioning.
  Maximum Activity Score (MAS) is highest item number answered still doing. Represents highest oxygen demanding activity that respondent still performs.
  Adjusted Activity Score (AAS) is MAS minus total number of stopped doing responses below MAS. A measure of usual daily activities.
  Modified AAS is MAS minus total number of stopped doing responses below MAS but not penalized for not doing activities not permitted post transplant. The following items are not counted against the score:11,15,19,20,22,25,34,41,42,47,49,50,52,53,54,57,72,73,77,78.
Time Frame: baseline
Population: Only baseline surveys analyzed. Only 7 patients completed surveys at 6mo, not analyzed due to low number.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
units on a scale
  maximum activity score | 66 [6 to 87]
  adjusted activity score | 57 [2 to 82]
  modified adjusted activity score | 60 [2 to 82]

15. Secondary Outcome: Symptoms as Measured by Patient Self-report--Lee Chronic GVHD Symptom Scale
Description: Lee symptom scale (LSS) has subscales with min=0, max=100; results given are 12mo scores, with higher numbers indicating higher symptom burden.
Time Frame: baseline
Population: Only baseline surveys analyzed. Only 7 patients completed surveys at 6mo, not analyzed due to low number.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Carfilzomib)
Number analyzed (Participants) | 20
units on a scale
  skin scale | 32.5 [0 to 100]
  energy scale | 42.9 [7.1 to 96.4]
  lung scale | 5 [0 to 30]
  eye scale | 62.5 [0 to 100]
  nutrition scale | 5 [0 to 20]
  psychological scale | 25 [0 to 66.7]
  mouth scale | 0 [0 to 75]
  overall summary score | 21.6 [8.2 to 49.3]

ADVERSE EVENTS:
Time Frame: 30 days after stopping study drug
Arm/Group | Treatment (Carfilzomib)
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Carfilzomib) (N=20)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sepsis (Infections and infestations) | 2 (2)
fever/infusion reaction (General disorders) | 1 (1)
leg ulcers (Skin and subcutaneous tissue disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
acute renal failure/sepsis (Renal and urinary disorders) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nausea/vomitting/diarrhea (Gastrointestinal disorders) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Carfilzomib) (N=20)
bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
fungal lung infection (Infections and infestations) | 1 (1)
decreased lymphocyte count (Blood and lymphatic system disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1)
esophageal varices (Gastrointestinal disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
increased ALT (Hepatobiliary disorders) | 1 (2)
intermittent hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Left hip hemiarthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1)
myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
rhinovirus (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT02491359/Prot_SAP_000.pdf